CLINICAL TRIAL: NCT00052156
Title: A Phase III Randomized Double-Blind Pivotal Trial of Immunotherapy With a Polyvalent Melanoma Vaccine, CancerVax™ Vaccine Plus BCG Versus Placebo Plus BCG as a Post-Surgical Treatment for Stage IV Melanoma
Brief Title: Vaccine Therapy for Patients With Stage IV Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CancerVax Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV-MMAIT-4-001; JWCI-MC-4-001; NCT00003722 (obsolete NCT alias)
Record Dates: First submitted 2003-01-23; First posted 2003-01-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-04

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Canvaxin

INTERVENTIONS:
Biological: CancerVax vaccine (CANVAXIN)

SUMMARY:
This is a Phase III study in patients with melanoma that has spread to the lymph nodes and/or a distant organ, and who have had all of their cancer surgically removed. The purpose of this study is to evaluate the ability of the CancerVax™ vaccine to prevent or slow the recurrence of melanoma.

ELIGIBILITY:
* Must have Stage IV melanoma
* Must have had all clinically-detectable disease surgically removed
* Cannot be taking any medications, or undergoing any therapies which compromise the functioning of your immune system (ie. Some corticosteroids, and certain types of radiation therapy)
* Cannot have HIV or Hepatitis A, B, or C

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670

CONTACTS AND LOCATIONS:
Locations (77):
- United States (51):
  - Arizona Cancer Center, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Medical Group, Anaheim, California
  - Cedars Sinai Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Comprehensive Cancer Center at DRMC, Palm Springs, California
  - Kaiser Permanente Medical Group, Riverside, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Sharp Hospital, San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Mt. Sinai Comprehensive Cancer Center, Miami, Florida
  - University of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - The Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - OSF Saint Francis Medica Center, Peoria, Illinois
  - Wagner and Associates, Indianapolis, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - St. Agnes Healthcare, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center, Lutherville, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Spectrum Health - Butterworth Campus, Grand Rapids, Michigan
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - The Cancer Cener at Hackensack University Medical Center, Hackensack, New Jersey
  - Medical Center of Princeton, Princeton, New Jersey
  - Millard Fillmore Hospital, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Suny Health Science Center at Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Dayton Clinical Oncology Group, Dayton, Ohio
  - St. Lukes Hospital Cancer Center, Bethlehem, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - UT Southwest Medical Center- Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Health Care- Mckay-Dee Hospital, Ogden, Utah
  - Intermountain Health Care-LDS Hospital, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (6):
  - Royal Prince Alfred Hospital, Sydney, Sydney, New South Wales
  - NSW Breast Cancer Institute, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Brazil (2):
  - INCA (National Cancer Institute), Rio de Janeiro
  - Hospital Sirio Lebanes, São Paulo
- McGill University, Montreal, Quebec, Canada
- CHU Pitie-Salpetriere, Paris, France
- Germany (7):
  - Klinikum Augsburg, Augsburg
  - Charite- University Medicine, Berlin
  - University of Jena, Jena
  - University Hospial of Mannheim, Mannheim
  - University of Tuebingen, Tübingen
  - University of Ulm, Ulm
  - University Hospital Wuerzburg, Würzburg
- Cork University, Cork, Ireland
- Tel-Aviv Medical Center, Tel Aviv, Israel
- Italy (3):
  - Istituto Nazionale Tumori di Milano, Milan, Milan
  - Instituto Eurepeo di Oncologia, Milan, Milan
  - Istituto Nazionale dei Tumori, Naples
- University Hospital of Groningen, Groningen, Netherlands
- North Shore Hospital, Auckland, Auckland, New Zealand
- University of Zurich, Zurich, Switzerland
- Harley Street Clinic, London, England, United Kingdom

REFERENCES:
- [Derived] Faries MB, Mozzillo N, Kashani-Sabet M, Thompson JF, Kelley MC, DeConti RC, Lee JE, Huth JF, Wagner J, Dalgleish A, Pertschuk D, Nardo C, Stern S, Elashoff R, Gammon G, Morton DL; MMAIT-IV Clinical Trial Group. Long-Term Survival after Complete Surgical Resection and Adjuvant Immunotherapy for Distant Melanoma Metastases. Ann Surg Oncol. 2017 Dec;24(13):3991-4000. doi: 10.1245/s10434-017-6072-3. Epub 2017 Oct 10. PMID 29019177
- [Derived] Hoshimoto S, Faries MB, Morton DL, Shingai T, Kuo C, Wang HJ, Elashoff R, Mozzillo N, Kelley MC, Thompson JF, Lee JE, Hoon DS. Assessment of prognostic circulating tumor cells in a phase III trial of adjuvant immunotherapy after complete resection of stage IV melanoma. Ann Surg. 2012 Feb;255(2):357-62. doi: 10.1097/SLA.0b013e3182380f56. PMID 22202581
- See also: CancerVax Corporation Website — http://www.cancervax.com